Approval Number: 202210059DIPA

## National Taiwan University Hospital Clinical Trial Protocol

\* This protocol should include a "Clinical Trial Summary" on the cover page.

□Drug □Medical Device □Medical Technology Other: Purely Academic Research

## **I.Project Title**

Difference in aerosol-generating amount between wired magnetic-assisted capsule endoscopy system and esophagogastroduodenoscopy examination of varices in biliary atresia patients

## **II.Principal Investigator**

Dr. Jia-Feng Wu, Attending Physician / Professor

## **III.Co-Principal Investigator**

Dr. Ping-Huei Tseng, Attending Physician / Professor

Dr. Chi-San Tai, Attending Physician / Lecturer

## **IV.Specific Aims**

The goal of this clinical trial is to compare the safeness and effectiveness of traditional esophagogastroduodenoscope (EGD) and wired magnetically assisted capsule endoscopy (MACE) in the diagnosis of esophageal varices in biliary atresia (BA) patients.

#### V.English Abstract

**Background and aims:** Biliary atresia (BA) is the leading cause of chronic liver insufficiency, liver cirrhosis, esophageal varices, and liver transplantation in the world. Regular endoscope examination with prompt adjustment of therapeutic agents is key to avoid the occurrence of esophageal varices bleeding. During the pandemic of COVID-19, to offer a regular and safe endoscopy survey of esophageal varices in BA patients become a medical challenge issue in the world.

Our study aim to investigate the diagnostic utility and safety of a Magnetically Assisted Capsule Endoscopy (MACE) system as comparing with traditional esophagogastroduodenoscope (EGD) in BA patients for the esophageal varices survey. We also aim to clarify whether the MACE is a less aerosol -generating procedure than EGD during the survey of esophageal varices, and decrease the risk of SARS-CoV 2 transmission.

**Methods:** This is an open-labeled un-blind trail. We intend to include 25 BA patients > 6 years of age agree to receive MACE examination into the study group, and another 25 BA patients > 6 years of age

Approval Number: 202210059DIPA

who will receive regular EGD into the control group. After the signature of the inform consent, they will enter this study. During the examination, a DR-528 Handheld Particle Counter (Met One Instruments, Inc., Grants Pass, OR) will be applied to detect aerosol generated during the examination. The compliance, diagnostic accuracy, and safety between study and control groups will be analyzed.

Scientific merits and anticipated results: The MACE was approved to achieve similar diagnostic accuracy and safety as EGD in adult population in Taiwan. Since subjects receiving MACE examination may close their mouth and have a face mask during the procedure, we intend to prove the MACE is an efficient, safe and less aerosol-generating procedure than EGD in BA patients this study. With the results of this study, we may offer the evidence of a safe and efficient examination during the pandemic of COVID-19 to protect the patients and medical staffs.

#### VI.Background Introduction & Significance

**Research Purpose:** Our study aims to investigate the diagnostic utility and safety of the Magnetically Assisted Capsule Endoscopy (MACE) system compared to traditional esophagogastroduodenoscopy (EGD) in the surveillance of esophageal varices in patients with biliary atresia (BA). Additionally, we seek to determine whether MACE generates fewer aerosols than EGD during the examination, thereby potentially reducing the risk of SARS-CoV-2 transmission.

General Background Information: Biliary atresia (BA) is one of the leading causes of chronic liver failure, liver cirrhosis, esophageal varices, and the need for liver transplantation during childhood worldwide (1-4). Statistically, approximately 50% of patients with BA develop portal hypertension, and 26.5% are at risk of gastrointestinal variceal bleeding (5-7). Esophageal variceal bleeding often results in significant complications and risks. In adult patients with chronic hepatitis, clinical indicators such as APRI, FIB-4, Extended BAVENO, or BAVENO VI are commonly used to help predict the presence of significant esophageal varices (8, 9). However, previous studies in BA patients have shown that these clinical indicators are not accurate in predicting the risk of esophageal varices in this population. Therefore, in clinical practice, physicians still rely on invasive esophagogastroduodenoscopy (EGD) to diagnose and assess the severity of esophageal varices. Based on the severity of the esophageal varices, physicians adjust medication dosages to reduce the risk of unexpected variceal bleeding and its associated complications.

Since the outbreak of SARS-CoV-2 in Wuhan, China in 2019, COVID-19 has continued to spread widely across the globe and has been confirmed as a direct contact and droplet infection disease. As of

Approval Number: 202210059DIPA

June 2022, COVID-19 has resulted in nearly 541 million infections and over 6.3 million deaths worldwide. In Taiwan, it has caused 3.44 million infections and more than 6,000 deaths. Consequently, the pandemic has placed enormous pressure and strain on global healthcare systems. During the outbreak in Europe in 2021, it was reported that over 20% of healthcare workers in northern Italy were infected, severely disrupting normal medical operations and preventing patients with chronic illnesses from receiving necessary medical care (10).

Since conventional esophagogastroduodenoscopy (EGD) has been confirmed as a respiratory droplet-generating medical procedure (11), healthcare workers performing EGD during the COVID-19 pandemic are at risk of being exposed to patient infections during the examination (12). In response, international medical societies have developed guidelines recommending appropriate personal protective equipment (PPE) for endoscopists, pre-procedural COVID-19 screening, requirements for the endoscopic environment, and prioritization criteria for urgent versus elective endoscopic procedures during the pandemic (13-20). Elective and surveillance EGDs were often recommended to be postponed or deferred. During the pandemic in Taiwan, limitations in hospital bed availability, healthcare workforce shortages, and patient anxiety also led to the postponement or deferral of many routine endoscopic examinations. However, in patients with biliary atresia (BA), regular endoscopic surveillance and appropriate medical adjustment have been validated as crucial strategies to prevent unexpected esophageal variceal bleeding (21). Delaying routine endoscopic surveillance and medical interventions in BA patients may increase the risk of unexpected variceal bleeding and life-threatening events. In addition, during periods of severe COVID-19 outbreaks, patients often hesitated or declined routine medical examinations, further leading to disease progression and deterioration.

Therefore, how to balance the medical needs of patients with biliary atresia (BA) and ensure that they receive necessary endoscopic examinations during the pandemic, while protecting both patients and endoscopy personnel from COVID-19 infection to maintain the proper functioning of healthcare systems, has become an important medical issue. Magnetic-assisted capsule endoscopy (MACE) is a novel design that utilizes a disposable, externally magnetically controlled capsule connected by a tether to guide its movement through the gastrointestinal tract (22, 23). Previous studies conducted in Taiwan have already demonstrated the safety and diagnostic accuracy of MACE for upper gastrointestinal examinations (22, 23), while also avoiding the risks associated with anesthesia. Although MACE requires swallowing a tether, its invasiveness remains significantly lower than that of conventional endoscopy. Preliminary studies have shown favorable safety and patient acceptance (22, 23). During the examination, the patient swallows the capsule similarly to taking a pill, and can keep their lips closed and wear a mask throughout the procedure.

#### Approval Number: 202210059DIPA

This study aims to evaluate whether MACE can achieve diagnostic performance comparable to traditional EGD in detecting esophageal varices in BA patients, while reducing aerosol generation during the procedure, thereby protecting both patients and endoscopy personnel from the risk of SARS-CoV-2 infection.

#### VII.Reference

- (I.) Bezerra JA, Wells RG, Mack CL, Karpen SJ, Hoofnagle JH, Doo E, et al. BILIARY ATRESIA: Clinical and Research Challenges for the 21st Century. Hepatology. 2018 Sep;68(3):1163-1173.
- (II.) Hoofnagle JH. Biliary Atresia Research Consortium (BARC). Hepatology. 2004; 39: 891.
- (III.) Sokol RJ, Shepherd RW, Superina R, Bezerra JA, Robuck P, Hoofnagle JH. Screening and outcomes in biliary atresia: summary of a National Institutes of Health workshop. Hepatology. 2007; 46: 566-581.
- (IV.) Hartley JL, Davenport M, Kelly DA. Biliary atresia. Lancet. 2009; 374: 1704-1713.
- (V.) Sohn H, Park S, Kang Y, Koh H, Han SJ, Kim S. Predicting variceal bleeding in patients with biliary atresia. Scand J Gastroenterol. 2019 Nov;54(11):1385-1390.
- (VI.) Shneider BL, et al. Portal hypertension in children and young adults with biliary atresia. J Pediatr Gastroenterol Nutr. 2012;55(5):567
- (VII.) Lykavieris P, et al. Outcome in adulthood of biliary atresia: a study of 63 patients who survived for over 20 years with their native liver. Hepatology. 2005;41(2):366.
- (VIII.) Deng H, et al. Diagnostic Accuracy of APRI, AAR, FIB-4, FI, King, Lok, Forns, and FibroIndex Scores in Predicting the Presence of Esophageal Varices in Liver Cirrhosis, Medicine: October 2015 Volume 94 Issue 42 p e1795
- (IX.) Tafarel JR, et al. Prediction of esophageal varices in hepatic cirrhosis by noninvasive markers. Eur J Gastroenterol Hepatol. 2011 Sep;23(9):754-8. doi: 10.1097
- (X.) Humanitas University, Department of Biomedical Sciences, Rozzano (Milan). Italy.
- (XI.) Chan SM, Ma TW, Chong MKC, Chan DL, Ng EKW, Chiu PWY. A Proof of Concept Study: esophagogastroduodenoscopy Is an Aerosol-Generating Procedure and Continuous Oral Suction During the Procedure Reduces the Amount of Aerosol Generated. Gastroenterology 2020;159:1949–1951
- (XII.) Repici A, Pace F, Gabbiadini R, Colombo M, Hassan C, Dinelli M. Endoscopy Units and the Coronavirus Disease 2019 Outbreak: A Multicenter Experience From Italy. Gastroenterology 2020;159:363–366
- (XIII.) Tokar JL, et al. Updated AGA Recommendations on Pre-Endoscopy COVID-19 Testing. Gastroenterology 2021 May 21.
- (XIV.) Sultan S, Siddique SM, Altayar O, et al. AGA Institute Rapid Review and Recommendations on the Role of Pre-Procedure SARS-CoV-2 Testing and Endoscopy.

#### Approval Number: 202210059DIPA

Gastroenterology. 2020 Nov; 159(5): 1935–1948.e5.

- (XV.) British Society of Gastroenterology (BSG). Endoscopy activity and COVID-19: BSG and JAG guidance update 22.03.20. 2020
- (XVI.) Zhang Y, Zhang X, Liu L, Wang H, Zhao Q. Suggestions of Infection Prevention and Control in Digestive Endoscopy During Current 2019-nCoV Pneumonia Outbreak in Wuhan, Hubei Province, China. February 2020. 2020
- (XVII.) Soetikno R, Teoh AY, Kaltenbach T, et al. Considerations in performing endoscopy during the COVID-19 pandemic.
- (XVIII.) 2020 American Society for Gastrointestinal Endoscopy. Covid-19-asge-updates-for-members. 2020
- (XIX.) European Society for Gastrointestinal Endoscopy.

  ESGE-and-ESGENA-position-statement-on-gastrointestinal-endoscopy-and-the-covid-19-pandem ic. 2020
- (XX.) World Endoscopy Organisation (WEO). WEO recommendations on digestive endoscopy and the COVID-19 pandemic. 2020
- (XXI.) Lampela H, Kosola S, Koivusalo A, et al. Endoscopic Surveillance and Primary Prophylaxis Sclerotherapy of Esophageal Varices in Biliary Atresia. JPGN 2012;55: 574–579
- (XXII.) Lin YC, Chen CL, Kao YW, et al. Feasibility of Upper Gastrointestinal Examination in Home Care Setting with a Magnetically Assisted Capsule Endoscopy System: A Retrospective Study. Healthcare 2021, 9, 577.
- (XXIII.) Lien GS, Wu MS, Chen CN, Liu CW, Suk FM. Feasibility and safety of a novel magnetic-assisted capsule endoscope system in a preliminary examination for upper gastrointestinal tract. Surg Endosc 2017; DOI 10.1007/s00464-017-5887-0

#### **VIII.Experiment Designs & Methods**

(I.) Patient eligibility

A.Inclusion criteria:

- (A.) Biliary atresia patients > 6 years old
- (B.) Vital signs are stable
- (C.) Without acute gastrointestinal bleeding
- B. Exclusion Criteria:
  - (A.) Patients with metal implants, metal stent, artificial joints, bone plates, and bone screw
  - (B.) Patients with electronic devices, such as pacemakers, cochlear implants, or other

#### Approval Number: 202210059DIPA

implanted electronic medical devices

- (C.) Throat or esophageal obstruction leading to dysphagia patients
- (D.) Consciousness disturbance patients unable to swallow
- (E.) Patients with acute upper gastrointestinal bleeding
- (F.)Patients with platelet lower than 40K or PT INR > 1.5

#### (II.) Design of experiments:

A. Study Design: Prospective open-label trial.

#### B. Trial Procedure:

#### (A.) Endoscopic Examination

In this study, 25 patients aged 6 years or older with biliary atresia undergoing Magnetic-Assisted Capsule Endoscopy (MACE) for esophageal varices survey will be enrolled as the "study group," while another 25 patients aged 6 years or older with biliary atresia undergoing conventional esophagogastroduodenoscopy (EGD) for esophageal varices survey will be enrolled as the "control group."Both groups will prospectively enter the study after providing informed consent and signing the consent form. All patients will fast appropriately according to endoscopic examination guidelines before the procedure.Patients undergoing conventional EGD may choose to receive conscious sedation based on clinical needs.Patients undergoing MACE will be advised to keep their lips closed and wear a surgical mask during the examination. We will compare clinical parameters between the two groups, including examination completion rate, pain perception during the procedure, safety, and willingness to undergo the same examination again in the future.

#### (B.) Droplet Particle Measurement

During examinations in both the "study group" and the "control group," we will use the MET ONE airborne particle counter [DR-528 Handheld Particle Counter (Met One Instruments, Inc., Grants Pass, OR)], placed on a platform at the same horizontal level as the patient lying flat, to simultaneously measure the number of droplet particles generated during the procedure. We will then compare the differences in droplet particle counts between the two groups. The primary endpoint of this study is to analyze the

#### Approval Number: 202210059DIPA

difference in the number of droplet particles generated during the examinations between the "study group" and the "control group."The secondary endpoints are to analyze the examination completion rate, pain perception during the procedure, safety, and willingness to undergo the same examination again between the two groups.

(C.) Project Period: 11/01/2022-12/31/2026 (MM/DD/YYYY)

## IX.Required Medications or Medical Equipment and Quantities

- (I.) Magnetically Assisted Capsule Endoscopy (InsightEyes EGD): 50 sets
- (II.) Aries E500i Image Processor (including power cable) / Aries E500i (Model: FG-270-0008, Quantity: 1)
- (III.) InsightEyes Image Connector / InsightEyes EGD Dongle (Model: DG-001T, Quantity: 1): A connector that links the InsightEyes EGD to the image processor.
- (IV.)InsightEyes MFN Magnetic Controller / InsightEyes MFN (Model: FG-270-0001, Quantity: 1): A magnetic device used to manipulate and adjust the positioning angle of the InsightEyes EGD.



Stationary equipment: Arise E500i Image

Processor Medical-grade monitor (not
included in this product) InsightEyes Image

Connector

Controller: InsightEyes MFN Magnetic

Controller

Single-use medical devices: InsightEyes EGD

The above equipment has been approved by the Taiwan Food

and Drug Administration (TFDA) under Medical Device Permit No. 006509.

(V.)MET ONE airborne particle counter [DR-528 Handheld Particle Counter (Met One Instruments, Inc., Grants Pass, OR)]

**X.Format of medical record forms:** Study personnel will use separate case report forms (CRFs).

XI.Methods for Data Collection, Processing, Evaluation, and Statistical Analysis

Approval Number: 202210059DIPA

(I.) Collect and record the enrolled patients' basic information (including sex, age, height, weight, past medical history, and medication history), vital signs, pain index, blood test results within the past three months, and transient elastography values.

- (II.)Document the examination results of both the Magnetically Assisted Capsule Endoscopy (MACE) and conventional esophagogastroduodenoscopy (EGD), including the presence of esophageal varices and bleeding sites.
- (III.) Record the patients' acceptance of the examination and any adverse effects.
- (IV.)Record the particle count measurements obtained using the MET ONE Airborne Particle Counter [DR-528 Handheld Particle Counter (Met One Instruments, Inc., Grants Pass, OR)].

## XII.Statistical Analysis and Sample Size Calculation

We will analyze the results using STATA (version 17) and MedCalc (version 20) statistical software. Continuous variables will be analyzed using the Student t-test or Mann-Whitney U test to assess differences between the "study group" and the "control group." Categorical variables will be analyzed using the Chi-square or Fisher's exact test. A p-value of <0.05 will be considered the threshold for statistical significance. For the sample size calculation, we assume that the study group will wear surgical masks for the examination, which have an approximate filtration efficiency of 87-90%. Based on a 95% confidence interval and a 5% margin of error, we estimate that enrolling 50 subjects (25 in the study group and 25 in the control group) will provide sufficient power to detect statistically significant results.

#### **XIII.Adverse Reactions and Management**

To date, there have been no reported adverse events associated with the InsightEyes EGD wired magnetically controlled capsule endoscopy. In the event that the patient experiences choking, suffocation, or other adverse reactions during capsule ingestion, the physician will immediately discontinue the examination and retrieve the capsule endoscope.

# XIV.Principal Investigator and Co-Investigators' Academic and Professional Background, Publications, and Training

Please refer to the e-REC system for detailed information on the academic background, professional

Approval Number: 202210059DIPA

experience, publications, and training of the research personnel.

## XV. Responsibilities and Task List of Trial Personnel

| Title | Name | Responsibilities and Scope of Work |
|---|---|---|
| PI, Attending | Jia-Feng Wu | Study conception and execution, patient |
| Physician / Professor | | recruitment and assessment |
| Co-I, Attending | Ping-Huei Tseng | Study conception and execution, patient |
| Physician / Professor | recruitment and assessment | |
| Co-I, Attending | Chi-San Tai | Study conception and execution, patient |
| Physician / Lecturer | | recruitment and assessment |

#### **XVI.Subject Information and Informed Consent Form Format**

Please refer to the e-REC system for the subject informed consent form.

#### XVII.Preclinical data

None.

#### XVIII.Potential Physical and Psychological Risks and Benefits

None.

#### **XIX.Potential Financial Risks and Benefits**

Each participant will receive a nutritional supplement allowance of NT\$2,000.

#### **XX.**Conflict of Interest

None.

#### **XXI.Ownership of Research Outcomes**

The research outcomes will be jointly owned by the Principal Investigator and Insight Medical Solutions Co., Ltd.

#### **XXII.Funding Source**

This is an investigator-initiated study partially sponsored by the manufacturer.

#### **XXIII.Other Information**

None.

Approval Number: 202210059DIPA
Estimated Budget Table

| Item | Amount (NTD) | Description |
|---|---|---|
| Participant Transportation Fees | 100,000 | Transportation reimbursement |
| Research Nurse / Assistant | 682,000 | |
| Fees | | |
| Publication-Related Expenses | 50,000 | English editing and submission |
| | | fees |
| Hospital Administrative Fee | 30,000 | |
| Total | 862,000 | |